CLINICAL TRIAL: NCT06854510
Title: A Prospective, Single-Center, Randomized Controlled Study on Sodium Bicarbonate Mouthwash for the Prevention and Treatment of Radiation-Induced Oral Mucositis in Nasopharyngeal Carcinoma.
Brief Title: Sodium Bicarbonate for Reducing Radiation-Induced Oral Mucositis in Nasopharyngeal Carcinoma.
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ling-Long Tang, Prof., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2025-016-01
Record Dates: First submitted 2025-02-20; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Nasopharyngeal Cancinoma (NPC)
MeSH Terms: interventions — Mouthwashes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sodium Bicarbonate Solution Gargle Group (Experimental): Oral rinses using 2.5% sodium bicarbonate solution were administered daily throughout the radiotherapy course
  Interventions: Drug: Gargle with 2.5% sodium bicarbonate solution during radiotherapy
- Sodium Chloride Solution Gargle Group (Placebo Comparator): Oral rinses using 0.9% sodium chloride solution were administered daily throughout the radiotherapy course
  Interventions: Drug: Gargle with 0.9% sodium chloride solution during radiotherapy

INTERVENTIONS:
Drug: Gargle with 2.5% sodium bicarbonate solution during radiotherapy — In addition to routine oral care, patients received sodium bicarbonate solution gargle therapy from the initiation of radiotherapy until its completion. The treatment protocol is as follows:
  For patients with oral mucositis of grade 0 - 1, gargle with a 2.5% sodium bicarbonate solution (for 1 - 2 minutes each time) three times a day and spit out the liquid after each gargle. For patients with oral mucositis of grade ≥ 2, gargle with a 2.5% sodium bicarbonate solution (for 1 - 2 minutes each time) four to five times a day and spit out the liquid after each gargle.
  Arms: Sodium Bicarbonate Solution Gargle Group
Drug: Gargle with 0.9% sodium chloride solution during radiotherapy — In addition to routine oral care, patients received 0.9% sodium chloride solution gargle therapy from the initiation of radiotherapy until its completion. The treatment protocol is as follows: For patients with oral mucositis of grade 0 - 1, gargle with a 0.9% sodium chloride solution (for 1 - 2 minutes each time) three times a day and spit out the liquid after each gargle. For patients with oral mucositis of grade ≥ 2, gargle with a 0.9% sodium chloride solution (for 1 - 2 minutes each time) four to five times a day and spit out the liquid after each gargle.
  Arms: Sodium Chloride Solution Gargle Group

SUMMARY:
To evaluate whether the use of 2.5% sodium bicarbonate mouthwash throughout the entire course of radiotherapy for nasopharyngeal carcinoma reduces the severity of radiation-induced oral mucositis and improves patient adherence to treatment.

DETAILED DESCRIPTION:
With the improvement in the prognosis of locally advanced nasopharyngeal carcinoma (LA-NPC) patients, an increasing number of studys have turned their attention to the treatment-related toxicities in NPC patients. Common toxic reactions during the treatment of NPC patients include radiation-induced oral mucositis, radiation-induced skin injury, dysphagia, xerostomia, and hearing loss, etc. Among them, radiation - induced oral mucositis is one of the most common and severe complications during radiotherapy for NPC patients. More than half of LA-NPC will experience grade 3 - 4 radiation-induced oral mucositis.

Current international guidelines, including those from NCCN, ESMO, and the Multinational Association of Supportive Care in Cancer (MASCC), provisionally endorse sodium bicarbonate mouthwash as an adjunctive measure for RIOM management. The proposed mechanisms involve pH modulation of the oral cavity, microbial load reduction, and anti-inflammatory effects. Specifically: 1) NCCN guidelines incorporate sodium bicarbonate into multi-agent regimens with analgesics/anesthetics; 2) ESMO emphasizes its prophylactic potential in targeted therapy-associated mucositis; 3) MASCC consensus acknowledges its role in maintaining oral hygiene. However, these recommendations carry low evidence grades, with all guidelines explicitly highlighting the paucity of robust clinical data to substantiate efficacy claims.

To address this critical evidence gap, our research team proposes a randomized controlled trial to evaluate the efficacy of sodium bicarbonate mouthwash in mitigating RIOM severity throughout radiotherapy for LA-NPC. Given the current lack of high - level research evidence, the results of future research are expected to further confirm the effectiveness of sodium bicarbonate mouthwash in relieving radiation-induced oral mucositis during radiotherapy for NPC patients, improve the quality of life of NPC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed nasopharyngeal carcinoma.
2. No evidence of distant metastasis (M0).
3. Scheduled to receive radical radiotherapy.
4. Karnofsky scale (KPS) > 70.
5. Age 18-70 years.
6. Capacity for independent oral rinse administration without dysphagia.

Exclusion Criteria:

1. Patients receiving non-platinum-based concurrent chemotherapy regimens.
2. Radiation fields encompassing level Ib lymph nodes.
3. History of pre-existing oral mucosal disorders or recurrent oral ulceration.
4. Prior radiotherapy history.
5. Severe coexisting illness.
6. Pregnancy or lactation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
The incidence of grade ≥2 oral mucositis | from radiotherapy commencement until 14 days post-radiotherapy
  Oral mucositis grade was evaluated using RTOG (Radiation Therapy Oncology Group) criteria, with intergroup differences analyzed by Chi-square test.

SECONDARY OUTCOMES:
The incidence of grade ≥3 oral mucositis | from radiotherapy commencement until 14 days post-radiotherapy
  Oral mucositis grade was evaluated using RTOG (Radiation Therapy Oncology Group) criteria, with intergroup differences analyzed by Chi-square test.
The incidence of grade ≥1 oral mucositis | from radiotherapy commencement until 14 days post-radiotherapy
  Oral mucositis grade was evaluated using RTOG (Radiation Therapy Oncology Group) criteria, with intergroup differences analyzed by Chi-square test.
Oral fungal detection rate | from radiotherapy commencement until 14 days post-radiotherapy
  Fungal culture testing via oral swab should be performed when oral mucositis of grade ≥2 severity occurs.
Rate of oral pH decline | from radiotherapy commencement until 14 days post-radiotherapy
  Weekly electronic pH meter measurements were obtained pre-radiotherapy and during radiotherapy, with comparison of the decline rate from baseline to pH nadir.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No